CLINICAL TRIAL: NCT01311622
Title: An Open-Label, Single Centre Study to Assess the Pharmacokinetics and Pharmacodynamics of Warfarin When Co-Administered With Fostamatinib in Healthy Subjects
Brief Title: Effects of Administration of Fostamatinib on Blood Concentrations of Warfarin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00013
Record Dates: First submitted 2011-02-21; First posted 2011-03-09 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Rheumatoid Arthritis; Healthy Subjects
Keywords: drug-drug interaction; Phase 1; healthy subjects; warfarin; Rheumatoid arthritis; RA; fostamatinib open-label; pharmacokinetics; pharmacodynamics; level of Warfarin in the blood
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Warfarin; fostamatinib

ARMS (2):
- warfarin (Experimental)
  Interventions: Drug: warfarin
- warfarin and fostamatinib (Experimental)
  Interventions: Drug: warfarin; Drug: fostamatinib

INTERVENTIONS:
Drug: warfarin — 2 single 25 mg doses of Warfarin (5 x 5 mg tablets) administered 14 days apart
  Other Names: Marevan
Drug: fostamatinib — 2 x 50 mg Fostamatinib tablets (100 mg) twice daily for 13 days
  Arms: warfarin and fostamatinib

SUMMARY:
The purpose of this study is to determine whether fostamatinib influences the plasma concentration of warfarin and changes its blood thinning effect, and to investigate how safe and tolerable it is when administered with warfarin.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures (including genotyping screening sample for CYP2C9 and VKORC1).
* Males or females (of non-childbearing potential) aged 18 to 55 years (inclusive)
* Subjects must be negative for occult blood (stool card) prior to administration.
* Body weight of at least 50 kg and body mass index (BMI) between 18 and 35 kg/m2 inclusive

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may put the subject at risk because of participation in the study, or influence the results of the study.
* Healthy subject predicted to be most sensitive to warfarin based on CYP2C9 and VKORC1 genotypes.
* A protein C and/or protein S deficiency.
* Absolute neutrophil count of less than 2500/mm3 or 2.5 x 109/L
* Previous treatment with warfarin for a clinical indication (ie, participation in a previous warfarin interaction study is acceptable).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine PK parameters of R- and S-warfarin including but not limited to AUC and Cmax | From pre-dose to 168 h post dose relative to each single warfarin dose
  * Pharmacokinetics of warfarin measured by AUC
  * Pharmacokinetics of warfarin measured Cmax

SECONDARY OUTCOMES:
To measure International Normalised Ratio (INR) following administration of warfarin | From pre-dose to 168 h post dose relative to each single warfarin dose
To assess the steady-state pharmacokinetics of R406 (active metabolite of fostamatinib) by measuring AUCss, Cmax,ss, tmax,ss and CL/F | From predose on Day 11 until 12 h post dose on Day 14 relative to fostamatinib dosing
  * Steady state Pharmacokinetics of R406 measured by AUCss
  * Steady state Pharmacokinetics of R406 measured by Cmax
  * Steady state Pharmacokinetics of R406 measured by ss
  * Steady state Pharmacokinetics of R406 measured by tmax
  * Steady state Pharmacokinetics of R406 measured by CL/F
Safety and tolerability will be measured with regard to adverse events, laboratory assessments, vital signs, physical examination, and 12-lead ECG will be recorded. | From screening, Day -1 to Day 21 and follow up visit (Day 28)
  To examine the safety and tolerability of fostamatinib in combination with Warfarin: Adverse events, laboratory assessments, vital signs, physical examination, and 12-lead ECG

CONTACTS AND LOCATIONS:
Overall Officials: James Ritter, BM BCh MRCP FRCP, Principal Investigator — Quintiles, Phase 1 Unit, London; Mark Layton, MD MRCP (UK), Study Director — AstraZeneca
Locations (1):
- Research Site, London, United Kingdom